CLINICAL TRIAL: NCT03451526
Title: A Multi-centre Real-world Non-interventional Observational Study to Compare Prognoses of the Chinese Patients With N2 Non-small Cell Lung Cancer Who Received Adjuvant Chemotherapies and Perioperative Chemotherapies After Surgeries
Brief Title: A Study to Explore Prognoses of the Patients With N2 Non-small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Tang-Du Hospital (Other)
Collaborators: LinkDoc Technology (Beijing) Co. Ltd. (Industry)
Responsible Party: Principal Investigator, lixiaofei, Professor, Tang-Du Hospital
Other Study IDs: W-TONG04
Record Dates: First submitted 2018-02-02; First posted 2018-03-01 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Chinese; real-world evidences; NSCLC; surgeries
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgeries+adjuvant chemotherapies: Patients who received radical resection of lung cancer + adjuvant chemotherapies
  Interventions: Procedure: Surgeries
- Perioperative chemotherapies: Patients who received perioperative chemotherapies
  Interventions: Procedure: Surgeries

INTERVENTIONS:
Procedure: Surgeries — Surgeries plus adjuvant chemotherapies or perioperative chemotherapies
  Other Names: Adjuvant chemotherapies or perioperative chemotherapies

SUMMARY:
The trial was designed to compare the effectiveness of radical resections of lung cancer plus adjuvant chemotherapies and perioperative chemotherapies in the patients with N2 non-small cell lung cancer

DETAILED DESCRIPTION:
The trial is a multi-centre real-world non-interventional observational study. The Chinese patients with N2 non-small cell lung cancer enrolled from 2014 to 2017 who received radical resections of lung cancer and adjuvant chemotherapies will be included in the study and the study data on patient demographic/tumor biological characteristics and clinical treatment will be collected to evaluate compare effectiveness of radical resection of lung cancer plus adjuvant chemotherapies and perioperative chemotherapies after surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Patients with radical resection of lung cancer enrolled from 2014 to 2019;
* Pathologically diagnosed patients with non-small cell lung cancer;
* Patients with age > 18 years old;
* Patients who did not receive chest surgeries before hospitalization;
* Patients with N2 lymph nodes (+) after surgeries;
* Patients who received lymphadenectomy for one group or more groups of lymph nodes;

Exclusion Criteria:

* Patients with second primary tumors or multiple primary tumors;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pathologically diagnosed Chinese patients with N2 non-small cell lung cancer who received radical resection of lung cancer plus adjuvant chemotherapies and perioperative chemotherapies
Sampling Method: Non-Probability Sample
Enrollment: 2929 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Overall survival | 2014 - 2017
  Overall survival

SECONDARY OUTCOMES:
Disease-free survival | 2014 - 2017
  Disease-free survival

OTHER OUTCOMES:
Overall survivals in the subgroups | 2014 - 2017
  Overall survivals in the subgroups categorized by T staging
Disease-free survivals in the subgroups | 2014 - 2017
  Disease-free survivals in the subgroups categorized by T staging
Impact factors of overall survival as measured by age | 2014 - 2017
  Impact factors of overall survival as measured by age
Impact factors of overall survival as measured by gender | 2014 - 2017
  Impact factors of overall survival as measured by gender
Impact factors of overall survival as measured by BMI | 2014 - 2017
  Impact factors of overall survival as measured by BMI
Impact factors of overall survival as measured by tumor size | 2014 - 2017
  Impact factors of overall survival as measured by tumor size
Impact factors of overall survival as measured by tumor location | 2014 - 2017
  Impact factors of overall survival as measured by tumor location
Impact factors of overall survival as measured by T staging | 2014 - 2017
  Impact factors of overall survival as measured by T staging
Impact factors of overall survival as measured by clinical treatments | 2014 - 2017
  Impact factors of overall survival as measured by surgeries plus adjuvant chemotherapies and surgeries plus perioperative chemotherapies
Time to local recurrence | 2014 - 2017
  Time to local recurrence
Time to distant recurrence | 2014 - 2017
  Time to distant recurrence
Death rate within 30/90 days after surgeries | 2014 - 2017
  Death rate within 30/90 days after surgeries
Impact factors of death rate within 30/90 days after surgeries as measured by patient demographic characteristics | 2014 - 2017
  Impact factors of death rate within 30/90 days after surgeries as measured by patient demographic characteristics
Impact factors of death rate within 30/90 days after surgeries as measured by tumor biological characteristics | 2014 - 2017
  Impact factors of death rate within 30/90 days after surgeries as measured by tumor biological characteristics
Impact factors of death rate within 30/90 days after surgeries as measured by various modes of surgeries | 2014 - 2017
  Impact factors of death rate within 30/90 days after surgeries as measured by various modes of surgeries
Incidence of perioperative complications | 2014 - 2017
  Incidence of perioperative complications

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - China PLA General Hospital, Beijing, Beijing Municipality
  - Henan cancer hospital, Zhengzhou, Henan
  - Tongji Hospital Affiliated to Huazhong Technology Hospital, Wuhan, Hubei
  - Jiangsu cancer hospital, Nanjing, Jiangsu
  - Xi'an Tangdu Hospital, Xi'an, Shaanxi
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Huaxi Hospital Affiliated to Sichuan University, Chengdu, Sichuan
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - First Hospital Affiliated to Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No